CLINICAL TRIAL: NCT07144722
Title: Preliminary Evaluation of a Prehabilitation Program for Adults Awaiting Elective Heart Surgery and at Increased Risk of Postoperative Complications
Brief Title: Prehabilitation Program for Patients Awaiting Elective Heart Surgery at Increased Risk of Postoperative Complications: Feasibility and Potential Clinical Outcomes
Acronym: PRÉAD-CARDIAQU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Andre Denault, Anesthésiologiste, Montreal Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025-3527
Record Dates: First submitted 2025-08-02; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Surgery; Prehabilitation; Postoperative Complications
Keywords: exercise-based prehabilitation; pulmonary postoperative complications; teleprehabilitation; elective surgery; cardiac procedures
MeSH Terms: conditions — Postoperative Complications | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehab group (Experimental): Supervised by a physiotherapist, the program includes an initial functional assessment, individualized training (breathing exercises, aerobic and strengthening exercises), and weekly follow-up via videoconference or phone.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — What distinguishes this intervention from others is its hybrid delivery model, combining virtual more than in-person sessions to increase accessibility and adherence. Additionally, it incorporates specific inspiratory muscle training, which is often overlooked in standard prehabilitation programs, and emphasizes a personalized progression based on each participant's functional capacity and feedback. This tailored approach aims to optimize physical readiness before surgery while minimizing patient burden and travel requirements.
  Other Names: Inspiratory muscle training

SUMMARY:
The goal of this study is to learn if an exercise-based prehabilitation program can help people who are waiting for heart surgery and are at higher risk of complications recover better.

The main questions it aims to answer are:

Can a home-based prehabilitation program prescribed by a physiotherapist be done safely and realistically before heart surgery?

Participants will:

Take part in a personalized exercise program for a 8 to 16 weeks before surgery

Do breathing muscle training at home

Meet with a physiotherapist once a week, either in person or by video call

Be assessed before and after the program

Researchers will compare the postoperative results with those of patients who received usual care only.

ELIGIBILITY:
Inclusion Criteria:

* A high risk of perioperative and postoperative complications. This risk is determined based on the predictive thresholds for postoperative complications.
* A waiting period of at least 8 weeks.
* Access to a smartphone, tablet, or computer for videoconference visits.

Exclusion Criteria:

* Unstable angina, malignant arrhythmias, active endocarditis/myocarditis, myocardial infarction within the last 2 weeks, left main coronary artery disease ≥ 50% on coronary angiography, severe aortic stenosis, severe mitral insufficiency, and decompensated heart failure.
* Any other acute condition affecting vital signs or causing significant symptoms.
* Physical or cognitive impairment limiting the ability to participate in the program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate (%) | From enrollment to the end of treatment at maximum 16 weeks
  Proportion of eligible candidates who enroll in the study. Recruitment rate will be calculated as the number of participants enrolled divided by the number of eligible candidates, multiplied by 100.
Adherence Rate (%) | From enrollment to the end of treatment at maximum 16 weeks
  Proportion of participants who complete at least 70% of prescribed exercise sessions. Calculated as the number of participants meeting this threshold divided by the total number enrolled, multiplied by 100.
Program Safety - number of participants experiencing exercise-related adverse events | From enrollment to the end of treatment at maximum 16 weeks
  Count of participants experiencing one or more adverse events during the program, including angina, arrhythmias, myocardial infarction, acute heart failure, or sudden cardiac death of cardiac origin.
Participant Satisfaction - likelihood to recommend | From enrollment to the end of treatment at maximum 16 weeks
  Among participants who complete the program, the self-reported likelihood of recommending the program to others, measured on a numeric rating scale from 0 ("not at all likely") to 10 ("extremely likely").
Participant Satisfaction - likelihood to repeat | From enrollment to the end of treatment at maximum 16 weeks
  Among participants who complete the program, the self-reported likelihood of participating in the program again, measured on a numeric rating scale from 0 ("not at all likely") to 10 ("extremely likely").

SECONDARY OUTCOMES:
Maximal Inspiratory Pressure (cmH2O) | From enrollment to the end of treatment at maximum 16 weeks
  Difference between post-program and baseline values of maximal inspiratory pressure, measured in centimeters of water (cmH₂O) using a digital manometer.
Diaphragm Thickening Fraction (%) | From enrollment to the end of treatment at maximum 16 weeks
  Difference between post-program and baseline diaphragm thickening fraction, calculated as (thickness at end-inspiration - thickness at end-expiration) / thickness at end-expiration × 100 using ultrasound.
Grip Strength (kg) | From enrollment to the end of treatment at maximum 16 weeks
  Difference between post-program and baseline grip strength, measured in kilograms using a handheld dynamometer
5-repetition-sit-to-stand Test - Lower Limb Strength (seconds) | From enrollment to the end of treatment at maximum 16 weeks
  Difference between post-program and baseline time to complete five repetitions of the sit-to-stand test, measured in seconds.
5-meter Gait Speed (seconds) | From enrollment to the end of treatment at maximum 16 weeks
  Difference between post-program and baseline time to walk 5 meters, measured in seconds.
Functional Capacity - six-minute walk distance (meters) | From enrollment to the end of treatment at maximum 16 weeks
  Difference between post-program and baseline walking distance achieved in the Six-Minute Walk Test (6MWT), measured in meters
Number of participants with postoperative pulmonary complications | From the day of surgery through hospital discharge (average of 10 days)
  Count of participants with at least one postoperative pulmonary complication during hospital stay, as defined by clinical diagnosis documented in the medical record.
Duration of postoperative mechanical ventilation (hours) | From ICU admission after surgery until extubation (within hospital stay, average 24-72 hours)
  Time in hours from ICU admission to extubation
Recovery of Mobility - Postoperative day of first mobilization (day out of bed) | Un average of 1 - 3 days
  Postoperative day number on which the participant first sits out of bed.
Recovery of Mobility - Postoperative day of first ambulation | An average of 3 - 6 days
  Postoperative day number on which the participant first walks
Length of Postoperative Hospital Stay (days) | From the day of surgery through hospital discharge (average of 10 days)
  Number of days from the date of surgery to hospital discharge

OTHER OUTCOMES:
Postoperative pulmonary complication - Exploratory Outcome Measures - Comparison of Postoperative Recovery Indicators Between Study Participants and Historical Controls | The month following the completion of primary and secondary data collection
  Proportion (%) of participants, based on historical patient data from a sample of the same population as the study participants and from the year preceding the start of the project, who experienced at least one postoperative pulmonary complication. This will be recorded as described for the same variable in the secondary outcomes.
Postoperative Recovery - Exploratory Outcome Measures - Comparison of Postoperative Recovery - Duration of Mechanical Ventilation - Between Study Participants and Historical Controls | The month following the completion of primary and secondary data collection
  Duration of postoperative mechanical ventilation (hours) collected from historical patient records of the same population.
Postoperative Recovery - Exploratory Outcome Measures - Comparison of Postoperative Recovery - Recovery of mobility (first mobilization out of the bed) - Between Study Participants and Historical Controls | The month following the completion of primary and secondary data collection
  Postoperative day of first mobilization out of bed collected from historical patient records of the same population.
Postoperative Recovery - Exploratory Outcome Measures - Comparison of Postoperative Recovery - Recovery of mobility (first ambulation) - Between Study Participants and Historical Controls | The month following the completion of primary and secondary data collection
  Postoperative day of first ambulation collected from historical patient records of the same population.
Postoperative Recovery - Exploratory Outcome Measures - Comparison of Postoperative Recovery - Length of Hospital Stay - Between Study Participants and Historical Controls | The month following the completion of primary and secondary data collection
  Number of days from the date of surgery to hospital discharge collected from historical patient records of the same population.

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institut, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No